CLINICAL TRIAL: NCT05454319
Title: A Prospective Feasibility Study of Daily, Home-based Biofeedback Therapy Using Cerebri for Migraine Treatment.
Brief Title: Cerebri Biofeedback Feasibility Trial
Acronym: CER-MIG-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordic Brain Tech AS (Other Government)
Collaborators: St. Olavs Hospital (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 457654
Record Dates: First submitted 2022-07-01; First posted 2022-07-12 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Episodic Migraine
Keywords: Biofeedback
MeSH Terms: interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biofeedback Treatment Group (Experimental): Medical device
  Interventions: Device: Biofeedback

INTERVENTIONS:
Device: Biofeedback — Home-based biofeedback with medical device
  Other Names: CEREBRI

SUMMARY:
The purpose of this study is to investigate feasibility, usability, safety, efficacy, and tolerability of Cerebri biofeedback treatment for adults with episodic migraine.

In the study, the app-based biofeedback treatment Cerebri for migraines in adults will be tested. By using biofeedback, bodily signals that are thought to be associated with migraines, are measured. During the treatment, one sensor is attached on the shoulder to measure activity in the shoulder and neck muscles and one sensor is attached to the index finger to measure temperature and heart rate variability. By getting on-screen feedback on the phone, the user can learn techniques to reduce muscle tension, and increase finger temperature and heart rate variability. Reduced muscle tension, as well as increase in finger temperature and heart rate variability is a sign of relaxation and a deactivation of the nervous system, which can lead to fewer and less serious migraine attacks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, at the time of signing the informed consent
* Episodic migraines with or without aura diagnosed by a neurologist/physician per International Classification of Headache Disorders 3rd edition (ICHD-3).
* Having kept a headache diary with at least 80% adherence as part of routine clinical care in the last 28-days prior to inclusion.
* History of at least 4 and up to 14 days of migraines per 28-day period in the 3 months prior to screening, as recalled by the subject and confirmed in the clinical diary.
* At least three months of experience with smartphone and access to an iOS or Android phone at home.
* Capable of giving signed informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Onset of migraine before age 50 years.

Exclusion Criteria:

* Having a continuous background headache that never disappears completely.
* More than 14 days of headache (all types) per 28-day period.
* Subjects diagnosed with trigeminal autonomic cephalalgias and neuralgias.
* Subjects with secondary headache conditions.
* Subjects with headaches attributed by the treating neurologist/physician as being medication overuse headache according to the ICHD-3.
* Subject with pathologies that inhibit use of the device according to the instructions for use (e.g., blindness, deafness).
* Use of any concurrent preventive treatment (medications, meditation, physical therapy and psychotherapy as a headache treatment, acupuncture, etc.).
* Subjects who have previously failed three prophylactic pharmacological treatments.
* Subjects taking opioids (>3 days per month) or barbiturates at the time of screening.
* Subject participates in another clinical investigation.
* Alcohol overuse according to ICD-10-CM Code F10.1 or illicit drug use.
* Subject who is unlikely to follow Clinical Investigation Plan or where treatment seems futile in the opinion of the Investigator or have demonstrated an inability to sufficiently adhere to headache diary entries (<80%).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention assessed by number of days with logged headache per 28-day period, number of biofeedback sessions per 28-day period, and mean session duration | 3 months
  Extraction of data from headache diary and completed biofeedback sessions

SECONDARY OUTCOMES:
Usability of intervention assessed by mHealth app usability questionnaire (MAUQ) | 3 months
  Mean mHealth app usability questionnaire (MAUQ) score at treatment week 1 and 12
Usability of intervention assessed by modified System Usability Scale (SUS) questionnaire | 3 months
  Modified System Usability Scale (SUS) questionnaire score at treatment weeks 1 and 12
Initial estimates of efficacy and onset of efficacy assessed by number of migraine days | 3 months
  Change in the mean number of 28-day period migraine days from before treatment, to treatment weeks 1-4, weeks 5-8 and weeks 9-12.
Descriptive assessment of patients' belief about treatment efficacy assessed by Patient Global Impression of Change Scale (PGIC) | 3 months
  Change in self-reported treatment efficacy by the Patient Global Impression of Change Scale (PGIC) from before treatment to end-of-treatment
Change in subject-reported, headache-related disability assessed by Migraine-Specific Quality of Life Questionnaire version 2.1 (MSQ v2.1) | 3 months
  Change in subject-reported, headache-related disability measured using the Migraine-Specific Quality of Life Questionnaire version 2.1 (MSQv2.1), from before treatment to end-of-treatment
Descriptive assessment of users' experience of use of intervention, by semi-structured interviews to evaluate design and ease of use | 3 months
  Semi-structured interviews to evaluate design and ease of use of intervention, at treatment week 6 and 12, in a subset of subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Tore W Meisingset, MD, PhD, Principal Investigator — St. Olavs Hospital
Locations (1):
- St.Olavs Hospital HF, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided